CLINICAL TRIAL: NCT03255018
Title: Phase 2 Trial of Pembrolizumab in Relapsed and Refractory Gray-Zone Lymphoma (GZL), Primary Central Nervous System Lymphoma (PCNSL), and Other Extranodal Diffuse Large B-cell Lymphomas
Brief Title: Pembrolizumab in Relapsed and Refractory Gray-Zone Lymphoma (GZL), Primary Central Nervous System Lymphoma (PCNSL), and Other Extranodal Diffuse Large B-cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Roschewski, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170149; 17-C-0149
Record Dates: First submitted 2017-08-18; First posted 2017-08-21 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Non-Hodgkin Lymphoma; Lymphoma; Diffuse Large B-Cell Lymphoma; Gray-zone Lymphoma; Primary Central Nervous System Lymphoma
Keywords: Monoclonal Antibody; PD-1 Receptor
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with Gray-zone Lymphoma (GZL) or Extranodal Diffuse Large B-cell Lymphomas (DLBCL) (Experimental): Participants with gray-zone lymphoma (GZL) or extranodal DLBCL relapsed from or refractory to prior therapy with an anthracycline-based regimen
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Administered intravenously (IV) at a fixed dose of 200 mg every 3 weeks until disease progression or unacceptable toxicity; treatment may continue indefinitely if clinical benefit with options for treatment interruption if responding disease and re-treatment upon relapse.
  Other Names: Keytruda

SUMMARY:
Background:

B-cell lymphoma is a cancer of white blood cells that are found in lymph nodes. Some kinds of these cancers, such as gray-zone and extra-nodal, are rare and often aggressive. They are usually resistant to current treatments. Researchers want to see if a drug called pembrolizumab may treat these types of lymphoma.

Objective:

To collect data to see if it may be effective to give pembrolizumab to people with certain types of rare, aggressive B-cell lymphomas.

Eligibility:

People ages 18 and older who have a B-cell lymphoma, including gray-zone lymphoma or extra-nodal lymphoma

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Scans. They will lie in a machine that takes images.

A tissue sample from a previous procedure will be tested.

The study will be done in 21-day cycles. During the study, participants:

Will repeat the screening tests.

Will get the study drug as an infusion into a vein over about 30 minutes.

Will have a cheek swab and/or saliva sample collected.

May have a bone marrow aspiration. A needle will be put into the hipbone, and a small amount of bone marrow will be taken out.

May have a lumbar puncture. If cerebrospinal fluid is collected, researchers will study it.

May have an eye exam.

May provide tissue samples.

May have tumor samples taken.

Participants will have a visit about 30 days after the last dose of the study drug. They will then have 4 visits in year 1, 2 visits a year in years 2-5, and once each year thereafter. They will also be contacted by phone.

DETAILED DESCRIPTION:
Background:

* Gray-zone lymphomas (GZL) are rare, aggressive lymphomas that share clinical and biological features of diffuse large B-cell lymphoma (DLBCL) and Hodgkin lymphoma
* Standard upfront therapy for GZL is dose-intensive chemotherapy, though disease is often resistant; consolidative radiation therapy reserved for patients who are relapsed or refractory, and patients who fail radiation therapy have a poor prognosis
* Primary central nervous system lymphoma (PCNSL), primary testicular lymphoma (PTL), primary breast lymphoma (PBL), primary cutaneous DLBCL, leg-type, and intravascular B-cell lymphoma (IVBCL) are rare, aggressive extranodal subsets of DLBCL that usually have gene expression signatures of activated B-cell (ABC) DLBCL
* ABC-DLBCL has cure rates below 40% after standard therapy, and is associated with late recurrences, often involving the central nervous system (CNS) where treatment options are limited by chemotherapy resistance and an inability of many agents to cross the blood-brain barrier
* Molecular biology studies of GZL and extranodal DLBCL have identified potentially targetable genetic features involving the programmed death-1 (PD-1) signaling pathway
* A high proportion of GZL, PCNSL, and PTL cases have copy number alterations or chromosomal rearrangements involving the PD-1 ligands, programmed death-ligand 1 (PD-L1) and programmed death-ligand 2 (PD-L2)
* Pembrolizumab, a humanized immunoglobulin G4 (IgG4) monoclonal antibody that targets the PD-1 receptor, is a rational therapeutic target for patients with relapsed and refractory GZL, PCNSL, PTL, and other extranodal DLBCL

Objectives:

-To determine the best overall response rate of pembrolizumab in patients with relapsed and refractory GZL and extranodal DLBCL

Eligibility:

* Confirmed diagnosis of B-cell lymphoma, relapsed from or refractory to prior:

  * Cohort 1: B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and classical Hodgkin lymphoma (i.e., Gray-zone lymphoma or GZL)
  * Cohort 2: Extranodal diffuse large B-cell lymphoma involving one or more of the specified extranodal sites (i.e., extranodal DLBCL)
* Adequate bone marrow and organ function defined
* Age greater than or equal to 18 years

Design:

* Phase 2 study of patients with relapsed and refractory GZL and extranodal DLBCL
* Patients will be treated with pembrolizumab 200 mg (flat dose) intravenous (IV) every 3 weeks provided they have clinical benefit and no unacceptable toxicity; patients who achieve a complete response (CR) will have the option stop after 1 year of therapy.
* All responding patients (CR, partial response (PR), or stable disease (SD) with clinical benefit) who subsequently relapse or progress within 1 year after discontinuation of study drug are eligible for re-treatment.
* At least 20 evaluable patients each with GZL and DLBCL will be evaluated on this protocol for the primary endpoint (overall accrual ceiling of 52 patients)

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have a diagnosis of B-cell lymphoma confirmed by Laboratory of Pathology, National Cancer Institute (NCI), that is relapsed from or refractory to prior therapy as follows:

  * Cohort 1: B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and classical Hodgkin lymphoma (i.e., Gray-zone lymphoma or GZL)
  * Cohort 2: Extranodal diffuse large B-cell lymphoma involving one or more of the specified extranodal sites (i.e., extranodal diffuse large B-cell lymphoma (DLBCL). The following subtypes are included (they do not have to be confirmed as non-germinal center (non-GCB) subtype for study entry):

    * Primary central nervous system (CNS) lymphoma (PCNSL)
    * Primary testicular lymphoma (PTL)
    * Primary breast lymphoma (PBL)
    * Primary cutaneous DLBCL, leg-type
    * Intravascular large B-cell lymphoma (IVBCL)
    * Diffuse large B-cell, not otherwise specified (NOS), activated B-cell type, involving 1 or more extranodal site

NOTE: For GZL, diagnosis will be in accordance with the 2016 World Health Organization classification of lymphoid malignancies. Patients diagnosed with other extranodal DLBCL subtypes or that are not otherwise specified (NOS) must involve at least 1 extranodal site and must be considered non-GCB by local immunohistochemistry algorithms. Cases that are non-GCB by the Hans criteria are considered eligible as well as cases of DLBCL that are both cluster of differentiation 10 positive (CD10+) and multiple myeloma 1 positive (MUM1+).

* Evaluable disease by clinical exam (i.e., palpable lymphadenopathy, measurable skin lesions, etc.), laboratory assessment (i.e., lymphoma involvement of bone marrow or peripheral blood by morphology, cytology or flow cytometry), and/or imaging (measurable lymph nodes or masses on computed tomography (CT) or magnetic resonance imaging (MRI) and/or evaluable fluorine-18-deoxyglucose (FDG)-avid lesions on positron emission tomography (PET)
* Adequate tumor tissue (archival or fresh) must be available for correlative studies. NOTE: Tumor tissue may be from any previously collected tissue and adequacy is at the discretion of the Principal Investigator. If prior tissue is not available, patient must be willing to undergo baseline tumor biopsy.
* Be 18 years of age or older on day of signing informed consent
* Adequate performance status (PS) as follows:

  * Patients greater than or equal to 18 years must have Eastern Cooperative Oncology Group (ECOG) 0-1 (and Karnofsky greater than or equal to 60%)

NOTE: Patients greater than or equal to 18 years with an ECOG PS of 2 and Karnofsky greater than or equal to 60 will be considered eligible at the discretion of the Principal Investigator if decreased ECOG performance status is felt to be related to residual neurologic deficits caused by CNS disease involvement that are not progressive or anticipated to cause clinical management problems during study participation.

- Adequate organ function as evidenced by the following laboratory parameters (unless related to lymphoma infiltration at the discretion of the investigator):

* Absolute neutrophil count (ANC) greater than or equal to 750 /mcL
* Platelets greater than or equal to 50,000/mcL (transfusions not permitted)
* Hemoglobin greater than or equal to 9 g/dL (transfusions permitted)
* Serum creatinine: Adults: less than or equal to 1.5 times upper limit of normal (ULN). Children: age greater than or equal to 14: less than or equal to 1.5 mg/dL OR measured or calculated creatinine clearance (glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl):

Greater than or equal to 30 mL/min/1.73 m(2) for subject with creatinine levels > 1.5 times institutional ULN (CrCl should be calculated per institutional standard)

--Serum total bilirubin less than or equal to 1.5 times ULN

OR

Direct bilirubin less than or equal to ULN for patients with total bilirubin levels > 1.5 ULN

* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 times ULN (less than or equal to 5 X ULN if liver involvement)

  - The effects of pembrolizumab on the developing human fetus are unknown. For this reason, the following measures apply:
* Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the first dose of pembrolizumab.
* Men and women of childbearing potential (WOCBP) who are sexually active must agree to adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 120 days after the last dose of pembrolizumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participants must not be planning to conceive or father children within the projected duration of the trial, starting with the pre-screening/screening visit through 120 days after the last dose of pembrolizumab.
* WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

  * Ability of patient or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Patients with DLBCL who best fit the criteria of Epstein-Barr virus (EBV)+ DLBCL, NOS are not eligible
* Current or prior anti-cancer treatment prior to the first dose of pembrolizumab as defined below:

  * Chemotherapy, targeted small molecule therapy, or other anti-cancer treatment not otherwise specified below within 2 weeks
  * Radiation therapy within 2 weeks
  * Anti-cancer monoclonal antibody (mAb) treatment within 4 weeks
  * Use of an investigational agent (e.g., biologic, drug, or other) within 4 weeks
  * Allogeneic stem cell transplant within 100 days
  * Prior therapy with an anti-programmed cell death protein 1 (PD-1), anti-programmed death ligand 1 (PD-L1), or anti-programmed death ligand 2 (PD-L2) agent at any time
* No current use of systemic corticosteroids at physiologic doses > 10 mg/day of dexamethasone or equivalent are permitted. Patients receiving current systemic steroids must be on a stable steroid dose (i.e., less than or equal to 10 mg/day of dexamethasone or equivalent at the same dose for at least 7 days). Patients who recently discontinued systemic steroids must have completed them at least 7 days prior to entry.
* Uncontrolled intercurrent illness including, but not limited to the following that may limit interpretation of results or that could increase risk to the patient at the discretion of the investigator:

  * Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  * History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis; as well as active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV):

  ---Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV deoxyribonucleic acid (DNA) is undetectable.
  * Uncontrolled and/or symptomatic thyroid disease
  * Active graft-vs-host disease (GVHD) requiring treatment or any history of greater than or equal to grade II acute GVHD
  * Seizure activity within the past 4 weeks
  * Known mental or physical illness that would interfere with cooperation with the requirements of the trial or confound the results or interpretation of the results of the trial and, in the opinion of the treating investigator, would make the patient inappropriate for entry into the study.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab, breastfeeding must be discontinued if the mother is treated with pembrolizumab
* Received a live vaccine within 30 days of planned start of study therapy. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab unless felt to be in the best interests of the patient in the opinion of the investigator
* Known additional malignancy that requires active systemic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All large-scale genomic sequencing data will be shared with subscribers to the Database of Genotype and Phenotype (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the Database of Genotype and Phenotype (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0149.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 Gray-Zone Lymphoma (GZL): Cohort 1: B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and classical Hodgkin lymphoma (i.e., Gray-zone lymphoma or GZL)
  Participants will be treated with pembrolizumab 200 mg (flat dose) intravenous (IV) every 3 weeks provided they have clinical benefit and no unacceptable toxicity; participants who achieve a complete response (CR) will have the option to stop after 1 year of therapy.
- Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL): Cohort 2: Extra-nodal diffuse large B-cell lymphoma involving one or more of the specified extra-nodal sites (i.e., extra-nodal DLBCL)
  Participants will be treated with pembrolizumab 200 mg (flat dose) intravenous (IV) every 3 weeks provided they have clinical benefit and no unacceptable toxicity; participants who achieve a complete response (CR) will have the option to stop after 1 year of therapy.
Period: Overall Study
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
Started | 2 | 10
Completed | 2 | 3
Not Completed | 0 | 7
Not completed — Death on study | 0 | 5
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data collected for one participant in the DLBCL cohort who withdrew consent is reported in the table.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL) | Total
Number analyzed (Participants) | 2 | 10 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 6 | 7
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.53 (25.26) | 65.06 (7.25) | 62.93 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 8 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 2 | 8 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 7 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 10 | 12
Baseline Programmed Death-Ligand 1 (PD-L1) Status [Count of Participants; unit: Participants] — Positive means that tumor cells stained positive for PD-L1 and negative means no staining was visible. This is done by histologic review by pathologists.
  Not all participant's received tumor cell analyses due to tissue availability. Population: No tissue available for analyses for one participant in Cohort 1 and 8 participants in Cohort 2.
  Participants
    Positive: number analyzed (Participants) | 1 | 2 | 3
    Positive | 0 | 1 | 1
    Negative: number analyzed (Participants) | 1 | 2 | 3
    Negative | 1 | 1 | 2
Baseline Bone Marrow Involvement [Count of Participants; unit: Participants] — Positive means that lymphoma cells were present in the bone marrow at baseline and negative means that no lymphoma was seen by histologic confirmation.
  Not all participant's received bone marrow biopsies since per protocol they were only done if clinically indicated. Population: No bone marrow biopsy performed for 5 participants in cohort 2.
  Participants
    Positive: number analyzed (Participants) | 2 | 5 | 7
    Positive | 0 | 1 | 1
    Negative: number analyzed (Participants) | 2 | 5 | 7
    Negative | 2 | 4 | 6
Baseline Cerebral Spinal Fluid (CSF) Involvement [Count of Participants; unit: Participants] — Positive means that lymphoma cells were detected in the CSF by flow cytometry. Negative means no lymphoma cells were detected by flow cytometry.
  Not all participant's received lumbar punctures with CSF analysis since per protocol they were only done if clinically indicated. Population: 2 participants did not receive lumbar punctures in Cohort 1 and Cohort 2.
  Participants
    Positive: number analyzed (Participants) | 0 | 8 | 8
    Positive | 0 | 4 | 4
    Negative: number analyzed (Participants) | 0 | 8 | 8
    Negative | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate of Pembrolizumab in Participants With Relapsed/Refractory Gray-zone Lymphomas (GZL) and Extra-nodal Diffuse Large B-cell Lymphomas (DLBCL)
Description: Response was assessed by the International Working Group (IWG) response criteria which utilizes computed tomography (CT) scan to measure lymph node masses to assess response, bone marrow biopsies and aspirates done only if positive at the time of diagnosis or if clinically indicated. Response is calculated by measuring the sum of the products of all target lesions and then calculating the percent change from baseline or nadir. Products are calculated by multiplying the longest length by the perpendicular width of each target lesion. Confirmed complete response is <1 cm lymph nodes/lymph node masses; unconfirmed complete response is >1 cm lymph nodes and >75% decrease in size of lymph node masses; partial response is ≥50% decrease in size of lymph nodes/lymph node masses; and progression is >50% new or increased lymph node masses/lymph nodes. Complete response (confirmed) followed by complete response(unconfirmed) and partial response are associated with better outcomes in that order.
Time Frame: Up to 24 months
Population: 9/10 participants are analyzed in the DLBCL cohort because 1 participant was not evaluable due to withdrawal of consent prior to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
Number analyzed (Participants) | 2 | 9
percentage of participants
  Complete Response | 50 | 0
  Unconfirmed Complete Response | 0 | 0
  Partial Response | 0 | 11
  Progressive Disease | 50 | 89

2. Secondary Outcome: Number of Grades 1-5 Adverse Events in Participant With Gray-zone Lymphomas (GZL) and Extra-nodal Diffuse Large B-cell Lymphomas (DLBCL)
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade 1 is mild. Grade 2 is moderate. Grade 3 is serious. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Adverse events are collected from the first dose of therapy through 30 days past the last dose of study drug or start of new anti-cancer therapy, approximately 5 months and 7 days for cohort 1, and 44 months and 25 days for cohort 2.
Population: 9/10 participants are analyzed in the DLBCL cohort because 1 participant enrolled in the DLBCL cohort was not evaluable due to withdrawal of consent prior to treatment.
Measure: Number; unit: adverse events
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
Number analyzed (Participants) | 2 | 9
adverse events
  Grade 1 | 5 | 35
  Grade 2 | 0 | 20
  Grade 3 | 0 | 8
  Grade 4 | 0 | 2
  Grade 5 | 0 | 0

3. Secondary Outcome: Best Overall Response Rate According to the 5-point Lugano Classification for Interpreting 18 F-fluorodeoxyglucose (FDG)-Positron Emission Tomography (PET) Scans
Description: The response rate is calculated by dividing the number of participants that had a complete response (CR) or partial response (PR) to therapy measured on positron emission tomography (PET) scan in accordance with the 5-point Lugano classification. Best overall response is the best response (complete or partial response) recorded from the start of the treatment until disease progression/recurrence. The 5-Point Scale Deauville criteria scores the most intense uptake in a site of initial disease: no uptake or no residual uptake, slight uptake, but above blood pool, uptake above mediastinal but below or =to uptake in liver, uptake slightly to moderately higher than liver, & markedly increased uptake. 5Point Scale ranges:1 to 5, 1=best; 5=worst: 1, no uptake above background; 2, uptake ≤ mediastinum; 3, uptake > mediastinum but ≤ liver; 4, uptake moderately > liver; 5, uptake markedly higher than liver; X. CR=scores 1-3 on & PR is calculated by measured change from baseline (score 4 or 5).
Time Frame: every 3-6 months for 24 months
Population: For this outcome only 1 out of the 2 participants in the GZL cohort had a PET scan at the time of best response. In the DLBCL cohort only 6 out of the 9 had a PET Scan at the time of best response.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
Number analyzed (Participants) | 1 | 6
percentage of participants
  Complete Response | 100 | 0
  Partial Response | 0 | 0
  Stable Disease | 0 | 0
  Progressive Disease | 0 | 100

4. Secondary Outcome: Duration of Response for Participants Who Respond to Pembrolizumab
Description: DOR is beginning at the date clinical response is first identified; measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is documented and will be estimated for each of the two types of lymphoma individually using Kaplan-Meier curves with appropriate confidence intervals reported. Response was assessed by the International Working Group response criteria (Cheson et al.). Complete response is <1 cm lymph nodes/lymph node masses, and normal bone marrow/physical exam (PE); unconfirmed complete response is >1 cm lymph nodes and >75% decrease lymph node masses, normal PE and indeterminate in bone marrow; partial response is ≥50% decrease in lymph nodes/lymph node masses, decrease in liver/spleen and irrelevant in bone marrow; and progression is >50% new or increased lymph node masses/lymph nodes, enlarging liver/spleen, and reappearance in bone marrow.
Time Frame: every 3-6 months for 24 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
Number analyzed (Participants) | 2 | 9
Months | 18.25 [0 to 36.5] | 0.9 [0 to 0.9]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, or death, whichever occurs first. PFS will be estimated for each of the two types of lymphoma individually using Kaplan-Meier curves with appropriate confidence intervals reported. Response was assessed by the International Working Group response criteria (Cheson et al.). Disease relapse is decline in prognosis and progression >50% increase in lymph node masses/lymph nodes, enlarging liver/spleen, new sites and reappearance in bone marrow.
Time Frame: up to 2 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
Number analyzed (Participants) | 2 | 9
Months | NA [NA to NA] — Median PFS not reached due to more than 50% of participants in the GZL cohort not experiencing a progression event. | 1.4 [0.5 to 2.3]

6. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, alternative therapy for lymphoma given (such as radiation), or death, whichever occurs first. EFS will be estimated for each of the two types of lymphoma individually using Kaplan-Meier curves with appropriate confidence intervals reported. Response was assessed by the International Working Group response criteria (Cheson et al.). Disease relapse is decline in prognosis and progression >50% increase in lymph node masses/lymph nodes, enlarging liver/spleen, new sites and reappearance in bone marrow.
Time Frame: up to 2 months
Population: 1 participant in the GZL cohort, and 1 participant enrolled in the DLBCL cohort 1 were not evaluable due to withdrawal of consent prior to treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
Number analyzed (Participants) | 2 | 9
Months | NA [NA to NA] — Median EFS not reached due to more than 50% of participants in the GZL cohort not experiencing a progression event. | 1.4 [0.5 to 2.3]

7. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from treatment start date until date of death from any cause, date last known alive or last follow up. OS will be estimated for each of the two types of lymphoma individually using Kaplan-Meier curves with appropriate confidence intervals reported.
Time Frame: every 3-6 months, up to 2.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
Number analyzed (Participants) | 2 | 9
Months | NA [NA to NA] — Median OS was not reached due to more than 50% of participants still being alive. | 28.8 [1.1 to NA] — The upper confidence interval (CI) is not estimable. The upper CI is not estimable when there are insufficient (or no) events past the time reported to calculate the upper CI limit. It is mathematically not possible to determine the upper limit in those cases.

8. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the participant or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse events are collected from the first dose of therapy through 30 days past the last dose of study drug or start of new anti-cancer therapy., approximately 5 months and 7 days for cohort 1, and 44 months and 25 days for cohort 2.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
Number analyzed (Participants) | 2 | 9
Participants | 2 | 9

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the first dose of therapy through 30 days past the last dose of study drug or start of new anti-cancer therapy., approximately 5 months and 7 days for cohort 1, and 44 months and 25 days for cohort 2.
Arm/Group | Cohort 1 Gray-Zone Lymphoma (GZL) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL)
All-Cause Mortality (participants affected / at risk) | 0/2 | 5/9
Serious Adverse Events (participants affected / at risk) | 0/2 | 5/9
Other Adverse Events (participants affected / at risk) | 2/2 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Gray-Zone Lymphoma (GZL) (N=2) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL) (N=9)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Eye disorders - Other, vision decreased (Eye disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Gray-Zone Lymphoma (GZL) (N=2) | Cohort 2 Extra-nodal Diffuse Large B-cell Lymphoma (DLBCL) (N=9)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysarthria (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (4)
Fever (General disorders) | 0 (0) | 1 (5)
Flatulence (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 3 (3)
Gastrointestinal disorders - Other, Thrush (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Pain (General disorders) | 0 (0) | 2 (3)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03255018/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03255018/ICF_001.pdf